CLINICAL TRIAL: NCT01012544
Title: The MAgnitude of Platelet Inhibition and the Pharmacokinetics of a 600 mg Loading Dose of Clopidogrel, in Different Patient CATegories (Stable Angina Versus Acute-coronary Syndromes Versus ST-elevated Myocardial Infarction).
Brief Title: Platelet Reactivity in Stent Thrombosis Patients
Acronym: MAPCAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, J.M. ten Berg, Cardiologist, MD, PhD, FESC, FACC, St. Antonius Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAPCAT01
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Stent Thrombosis
Keywords: clopidogrel; pharmacokinetics; platelet function tests; platelet reactivity
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stent thrombosis patients (Active Comparator): Patients with a history of a stent thrombosis
  Interventions: Drug: Clopidogrel
- Patients without a history of a stent thrombosis (Active Comparator): Patients without a history of stent thrombosis
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — both arms of the study (patients with a history of stent thrombosis as well as patients who did not suffer from a stent thrombosis) will be given a 600 mg loading dose of clopidogrel
  Other Names: Plavix

SUMMARY:
Recent studies have demonstrated a marked interindividual variability of clopidogrel's capacity to inhibit platelet aggregation with a substantial proportion (11-34%) of the patients considered non-responders to clopidogrel treatment. Variable intestinal absorption is suggested to contribute to the inconsistencies in response to clopidogrel. However, little is known about intestinal absorption in subjects who had suffered from a stent thrombosis. The MAPCAT-study has been designed to investigate whether plasma pharmacokinetics (represented by Cmax, Tmax and the AUC) after a 600 mg loading dose are significantly different between subjects who have suffered a stent thrombosis and subjects who have not suffered a stent thrombosis.

DETAILED DESCRIPTION:
Objectives:

The first objective of the MAPCAT-study is to investigate whether plasma pharmacokinetics (Cmax, Tmax and AUC) of an additional 600 mg loading dose are impaired in patients with a history of stent thrombosis.

The second objective of the MAPCAT study is to investigate whether genetic polymorphisms in receptors, enzymes and ligands involved in the process of thrombosis and haemostasis as well in the conversion-process of clopidogrel into its metabolites do have influence on both the absolute magnitude of platelet inhibition and Cmax, Tmax and AUC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of a stent thrombosis in the period 2004-2008.

Exclusion Criteria:

* Persistent acute ST-segment elevation
* Successful revascularization during the qualifying hospitalization, prior to study entry
* Acute pulmonary edema, hypotension, or evidence of cardiogenic shock
* Clinically significant liver disease
* End stage kidney disease requiring dialysis
* Use at study entry of drugs that are strong inhibitors of cytochrome P450 3A4 and CYP3A5 (i.e. clarithromycin, erythromycin, itraconazole, ketoconazole)
* Contraindications to antithrombotic/antiplatelet therapy
* Failed coronary intervention in the previous 2 weeks
* Malignancies
* Increased risk of bleeding (previous stroke in the past months, active bleeding or bleeding diathesis, recent trauma or major surgery in the last month, suspected aortic dissection, oral anticoagulation therapy with coumarin derivate within 7 days, recent use of GPIIb/IIIa inhibitors within 14 days, severe uncontrolled hypertension >180 mmHg unresponsive to therapy)
* Relevant hematologic deviations (haemoglobin <100g/L (6,2 mmol/L) or hematocrit <34%, platelet count <100 x 109 /L or platelet count > 600 x 109/L)
* Known allergy to clopidogrel
* Pregnancy (present or suspected)
* uncontrolled hypertension at time of randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of unchanged clopidogrel, its active thiol metabolite and its inactive carboxyl metabolite between the different patient groups after the administration of a 600 mg loading dose of clopidogrel. | 6 hours after the administration of a 600mg loading dose of clopidogrel

SECONDARY OUTCOMES:
The magnitude of platelet reactivity as measured with several commercial available platelet function tests before and 6 hours after the ingestion of the loading dose. | platelet reactivity measured at baseline and 6 hours after a 600 mg clopidogrel loading dose.
Exploratory Endpoint: prevalence of various genetic polymorphisms that might influence the pharmacokinetics of clopidogrel | blood obtained for genetic sampeling at timepoint of first study blood collection

CONTACTS AND LOCATIONS:
Overall Officials: J.M. ten Berg, MD, PhD, Principal Investigator — St Antonius center for platelet function research
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] Elsenberg EH, van Werkum JW, van de Wal RM, Zomer AC, Bouman HJ, Verheugt FW, Berg JM, Hackeng CM. The influence of clinical characteristics, laboratory and inflammatory markers on 'high on-treatment platelet reactivity' as measured with different platelet function tests. Thromb Haemost. 2009 Oct;102(4):719-27. doi: 10.1160/TH09-05-0285. PMID 19806258
- [Background] Taubert D, Bouman HJ, van Werkum JW. Cytochrome P-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 May 21;360(21):2249-50; author reply 2251. doi: 10.1056/NEJMc090391. No abstract available. PMID 19458375
- [Background] van Werkum JW, Heestermans AA, Zomer AC, Kelder JC, Suttorp MJ, Rensing BJ, Koolen JJ, Brueren BR, Dambrink JH, Hautvast RW, Verheugt FW, ten Berg JM. Predictors of coronary stent thrombosis: the Dutch Stent Thrombosis Registry. J Am Coll Cardiol. 2009 Apr 21;53(16):1399-409. doi: 10.1016/j.jacc.2008.12.055. PMID 19371823
- [Background] Heestermans AA, van Werkum JW, Schomig E, ten Berg JM, Taubert D. Clopidogrel resistance caused by a failure to metabolize clopidogrel into its metabolites. J Thromb Haemost. 2006 May;4(5):1143-5. doi: 10.1111/j.1538-7836.2006.01891.x. No abstract available. PMID 16689772
- [Background] Taubert D, von Beckerath N, Grimberg G, Lazar A, Jung N, Goeser T, Kastrati A, Schomig A, Schomig E. Impact of P-glycoprotein on clopidogrel absorption. Clin Pharmacol Ther. 2006 Nov;80(5):486-501. doi: 10.1016/j.clpt.2006.07.007. PMID 17112805
- [Derived] Bouman HJ, van Werkum JW, Breet NJ, ten Cate H, Hackeng CM, ten Berg JM. A case-control study on platelet reactivity in patients with coronary stent thrombosis. J Thromb Haemost. 2011 May;9(5):909-16. doi: 10.1111/j.1538-7836.2011.04255.x. PMID 21382172